CLINICAL TRIAL: NCT03723161
Title: Evaluation of the Ponto Bone Anchored Hearing System in a Pediatric Atresia Population
Status: Completed | Type: Observational
Sponsor: Oticon Medical (Industry)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: C64
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Hearing Loss; Conductive Hearing Loss; Atresia
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Conductive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment: Bone Anchored Hearing surgery using a BHX implant manufactured by Oticon Medical
  Interventions: Device: Bone Achored Hearing surgery

INTERVENTIONS:
Device: Bone Achored Hearing surgery — This is a observational study of pediatric patients undergoing bone anchored hearing surgery. The collected data will be used to assess the implant stability development of the Ponto BHX implant during up tp 24 months after implantation in a pediatric population undergoing bone anchored hearing surgery.

SUMMARY:
The purpose of this study is to in a proactive manner collect high quality data from a pediatric patients who have undergone a bone anchored hearing solution, using the Ponto BHX implant, in clinical practice. This to further increase the knowledge of using the system.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have decided to undergo a Bone Anchored Hearing Surgery
* Diagnosed with atresia
* Signed informed consent
* Patients between 2,5 - 18 years of age
* Patients eligible for one stage surgery

Exclusion Criteria:

* Not fluent in Swedish or English; subject and/or legal guardian
* Unwillingness to participate in follow up visits

Ages: 30 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients eligible for a bone anchored solution.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Stability 12 months | 12 months post surgery
  The development of implant stability during the first 12 months after implantation; as measured by difference in mean of (Implant Stability Quotient) ISQ low 12 months compared to surgery.

SECONDARY OUTCOMES:
Stability 24 months | 24 months post surgery
  Difference in mean of ISQ low at 24 months compared to surgery
Implant survival rate | 24 months post surgery
  Implant survival rate in percent compared to litterature
Performance audibility PTA4 | 1 month post surgery
  The difference between abutment-aided and softband-aided sound field Pure Tone Average of thresholds at frequencies 500, 1000, 2000 and 4000 Hz (PTA 4) in preoperative condition and at fitting.
Performance audibility | 1 month post surgery
  Difference between abutment-aided and softband-aided sound field Pure Tone thresholds at frequencies 500, 1000, 2000, 4000, 6000 and 8000 Hz) in preoperative condition and at fitting
Performance speech intelligibility | 1 month post surgery
  Difference between abutment-aided and softband-aided speech intelligibility in SNR in preoperative condition and at fitting.
Functional assessment | 12 months, 24 months
  Functional assessment as measured by change in Pediatric Evaluation of Aural/Oral Performance of Children (PEACH)
Skin conditions Holger | 7-10 days,12 months, 24 months post surgery
  Skin assessment as assessed with maximum Holgers score per patient. Maximum score 4. 0= no adverse skin reaction, 4=maximum adverse skin reaction.
Skin conditions IPS evaluation | 7-10 days,12 months, 24 months post surgery
  Skin condition as assessed by (Inflammation, Pain, Skin height/numbness (IPS) score. I scale randing from 0-4, Pain scale ranging from 0-2, Height scale ranging from 0-2. Total score 8, 0=no adverse skin reaction, 8=maximum adverse skin reaction
Sustainability of audibility PTA4 performance | 1 month, 12 months, 24 months post surgey
  Difference between abutment aided sound field PTA 4 over time
Sustainability of audibility performance | 1 month, 12 months, 24 months post surgey
  Difference between abutment aided sound field Pure Tone thresholds at frequencies 500, 1000, 2000, 4000, 6000 and 8000 Hz over time
Sustainability of speech intelligibility performance | 1 month, 12 months, 24 months post surgey
  Difference between abutment aided speech intelligibility over time

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No